CLINICAL TRIAL: NCT03540082
Title: Safe Landing Strategy in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17577
Record Dates: First submitted 2018-03-23; First posted 2018-05-30 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Fall Prevention; Fall Injury; Fall Safety
Keywords: Aging; Older Adults; Fall prevention; Fall safety; Safe landing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fall Exposure (Active Comparator): An instructor will implicitly be exposed to the falling technique. Each group will have 4 sessions to physically practice the skills with each practice session lasting about an hour.
  Interventions: Other: Fall Exposure
- Control (No Intervention): Written instructions will be provided on the correct way to fall without physical practice.
- Tuck and Roll Group (Other): An instructor will explicitly verbally and visually demonstrate the falling technique and provide feedback on participant performance. Each group will have 4 sessions to physically practice the skills with each practice session lasting about an hour.
  Interventions: Other: Tuck and Roll Group

INTERVENTIONS:
Other: Tuck and Roll Group — An instructor will explicitly verbally and visually demonstrate the falling technique and provide feedback on participant performance. Each group will have 4 sessions to physically practice the skills with each practice session lasting about an hour.
  Arms: Tuck and Roll Group
Other: Fall Exposure — An instructor will implicitly be exposed to the falling technique. Each group will have 4 sessions to physically practice the skills with each practice session lasting about an hour.
  Arms: Fall Exposure

SUMMARY:
The purposes of this project to examine whether older adults can learn safe landing strategy during a fall. The research hypotheses are three-fold: 1) To determine whether older adults can learn a safe landing strategy to reduce impact severity of falling; 2) To examine whether the training effect on the right side falls can be transferred to the left side falls; and 3) To examine 1-week and 3-month retention effect of fall strategy training in older adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30 kg/m2
* Healthy bone mass (2.5 SD of young)
* No tumbling experience

Exclusion Criteria:

* > 70 years old
* Bone fracture within 3 years
* Osteoporosis
* Blood thinners

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-19 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Safe Landing Strategy | 1-week and 3-months post
  To determine whether older adults can learn a safe landing strategy to reduce impact severity of falling through a composite outcome from the following measures:
  1. Forceplate measurements (CueFors2, Motek Medical)
  2. Motion capture (VICON, Oxford Metrics)
  3. Inertial sensor (BioStampRC, MC10)
  4. Short-term skill acquisition (Aim 1) will be quantified as change in hip impact force between baseline and post assessments on visit 4

SECONDARY OUTCOMES:
Retention effects | 3-months post
  Examine retention effect of fall strategy training through a composite score from the following:
  1. Participant questionnaire
  2. Track and review which participants attend all four study visits